CLINICAL TRIAL: NCT05121311
Title: Assessment of Neonatal Hyperbilirubinemia by NeoprediX B.1 Algorithm - Prospective Observational Study -
Brief Title: Assessment of Neonatal Hyperbilirubinemia by NeoprediX B.1 Algorithm
Acronym: Bili-PrediX1
Status: Completed | Type: Observational
Sponsor: NeoPredix AG (Industry)
Collaborators: Center for Pediatric Clinical Studies (CPCS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 507/2021B02
Record Dates: First submitted 2021-08-18; First posted 2021-11-16 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Newborn Jaundice
Keywords: newborn jaundice; Hyperbilirubinaemia
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborns under bilirubin monitoring: Bilirubin monitoring according to standard of care of the participating center
  Interventions: Diagnostic Test: NeoprediX B1 algorithm

INTERVENTIONS:
Diagnostic Test: NeoprediX B1 algorithm — Re-assessement of bilirubin measurements done according to standard of care of the participating center by the NeoprediX B1 algorithm

SUMMARY:
Due to actual standard of neonatal care bilirubin is monitored in neonates several times after birth to avoid hyperbilirubinemia. As the peak is often one or two days after discharge from hospital a more precise predication than the actual one is desirable to avoid needlessly follow-ups. The precision of an algorithm to predict bilirubin values 24-48h into the future is evaluated in this study.

DETAILED DESCRIPTION:
Neonatal jaundice is common and mostly transient without need for intervention. To identify infants at risk of bilirubin toxicity, bilirubin is measured several times after birth and before discharge home. As the peak bilirubin concentrations are reached at days 4-6 after birth, and most infants are discharged home around 48 hours after birth, parents are often asked to return to hospital one or two days after discharge with their newborn baby to have the bilirubin value checked in order to prevent that hyperbilirubinemia requiring treatment is not missed. A precise prediction of the course of bilirubin values based on the measurements done during the initial hospital stay after birth would be desirable to avoid unnecessary follow ups (both for the families and the health care system).

This study aims to evaluate the precision of the NeoprediX B1 algorithm. This algorithm predicts bilirubin values 24-48h into the future based on preceding values and some clinical variables. Five different scenarios will be explored, differing in the type, number and timepoints of measurements used for the prediction as well as the timepoint that is to be predicted.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infant
* gestational age at birth ≥ 34+0/7 weeks

Exclusion Criteria:

* Birth weight < 1500g
* Gestational age at birth > 42+6/7 weeks
* Genetically defined syndrome
* Severe congenital malformation adversely affecting life expectancy or admission for a priori planned palliative care
* Parents not fluent in German

Max Age: 72 Hours | Sex: All
Age Groups: Child
Study Population: Newborn infants
Sampling Method: Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Precision of predicted bilirubin value | 8 hours to 144 hours after birth
  Precision of the bilirubin value calculated by the NeoprediX B1 algorithm compared to the value measured by the center

CONTACTS AND LOCATIONS:
Overall Officials: Axel Franz, Prof., Principal Investigator — University Children's Hospital Tübingen
Locations (2):
- Germany (2):
  - KUNO Kinderklinik St. Hedwig, Regensburg
  - University Children's Hospital, Tübingen

IPD SHARING:
Plan to Share IPD: No